CLINICAL TRIAL: NCT06509659
Title: Methacholine Challenge Test (MCT) in Healthy Adults: Oscillometry Measured Alone Compared to Oscillometry and FEV1 During the Same Test
Brief Title: Methacholine Challenge Test (MCT) in Healthy Adults
Status: Recruiting | Type: Observational
Sponsor: Allergi- og Lungeklinikken, Elsinore (Network)
Responsible Party: Principal Investigator, Thomas Ringbæk, Principal Investigator, Allergi- og Lungeklinikken, Elsinore
Other Study IDs: Elsinore_Healthy
Record Dates: First submitted 2024-04-07; First posted 2024-07-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hyperreactive Airway Disease
Keywords: IOS; oscillometry; spirometry; bronchial hyperreactivity
MeSH Terms: conditions — Bronchial Hyperreactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy controls: No lung disease or symptoms. Negative methacholine Challenge Test.
  Interventions: Diagnostic Test: Methacholine Challenge Test

INTERVENTIONS:
Diagnostic Test: Methacholine Challenge Test — MCT with IOS alone versus MCT IOS and FEV1 combined
  Other Names: FEV1 measurement

SUMMARY:
Knowledge of Methacholine Challenge Test (MCT) and impedance Oscillometry (IOS) is limited. Only three studies have included adult patients, and none of these with healthy controls. The three studies have combined IOS and spirometry in the same test, although it is not recommended to perform IOS after a test that requires deep breathing, e.g. FEV1 measurement. Deep breathing is considered to affect the impedance via reduced tone in the smooth muscle.

DETAILED DESCRIPTION:
Asthma is a common chronic disease that is characterized by a history of variable respiratory symptoms and variable expiratory airflow limitation, and usually associated with airway hyperresponsiveness.

In general, FEV1 is used to test for airway hyperresponsiveness (AHR), and a 20% decrease after methacholine challenge test (MCT) is considered a positive test.

There is increasing recognition that the small airways are involved in 40-80% of patients with asthma, and the function of these airways is overlooked (the "silent zone") when measuring FEV1, which mainly reflects the function of the central airways.

Small airway dysfunction (SAD) can be assessed by IOS where pressure applied to the airways at a range of frequencies, and components of respiratory resistance and reactance are measured. Resistance at 5 Hz (R5) and 20 Hz (R20), respectively, represent total airway resistance and proximal airway resistance. The difference between these two values can be calculated (R5-R20). High R5-R20 and low reactance at 5 Hz (X5) indicate the presence of SAD.

Knowledge of MCT and IOS is limited. Only three studies have included adult patients, and none of these with healthy controls. These studies have combined IOS and spirometry in the same test, although it is not recommended to perform IOS after a test that requires deep breathing, e.g. FEV1 measurement. Deep breathing is considered to affect the impedance via reduced tone in the smooth muscle.

The investigators have the following objectives for these studies:

1. To determine the IOS response to MCT in healthy adults.
2. To investigate whether spirometry (FEV1) carried out in relation to MCT influences IOS by comparing the IOS response to MCT performed with and without spirometry in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Forced expiratory volume in the 1. second (FEV1) >80%
* FEV1/FVC-ratio >0,7
* FeNO <25 pbb
* Oxygen saturation (SatO2) >95%
* Negative methacholine Challenge Test = drop in FEV1 less than 20%

Exclusion Criteria:

* Any lung disease
* Lung symptoms
* Medicine for lung disease
* Tobacco smoking
* Ex-smokers with more than 5 package years
* BMI (body mass index) >40 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-23 (Estimated)

PRIMARY OUTCOMES:
Oscillometry; R5 | baseline (carried out with FEV1 measurement)
  Resistance at 5 Hz; kPa/L/s with FEV1 measurement
Oscillometry; R5 | 1-10 days from baseline and carried out without FEV1 measurement
  Resistance at 5 Hz; kPa/L/s change from baseline
Oscillometry; R20 | baseline (carried out without FEV1 measurement)
  Resistance at 20 Hz; kPa/l/s with FEV1 measurement
Oscillometry; R20 | 1-10 days from baseline and carried out without FEV1 measurement
  Resistance at 20 Hz; kPa/L/s change from baseline
Oscillometry; X5 | baseline (carried out without FEV1 measurement)
  Reactance at 5 Hz; kPa/l/s with FEV1 measurement
Oscillometry; X5 | 1-10 days from baseline and carried out without FEV1 measurement
  Reactance at 5 Hz; kPa/L/s change from baseline
Oscillometry; AX | baseline (carried out without FEV1 measurement)
  Area of reactance; kPa/L with FEV1 measurement
Oscillometry; AX | 1-10 days from baseline and carried out without FEV1 measurement
  Area of reactance; kPa/L change from baseline
Oscillometry; Fres | baseline (carried out without FEV1 measurement)
  Resonant frequency; Hz with FEV1 measurement
Oscillometry; Fres | 1-10 days from baseline and carried out without FEV1 measurement
  Resonant frequency; Hz change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Ringbæk, Principal Investigator — Allergy and Lung Clinic Elsinore
Locations (1):
- Thomas Ringbæk, Elsinore, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coates AL, Wanger J, Cockcroft DW, Culver BH; Bronchoprovocation Testing Task Force: Kai-Hakon Carlsen; Diamant Z, Gauvreau G, Hall GL, Hallstrand TS, Horvath I, de Jongh FHC, Joos G, Kaminsky DA, Laube BL, Leuppi JD, Sterk PJ. ERS technical standard on bronchial challenge testing: general considerations and performance of methacholine challenge tests. Eur Respir J. 2017 May 1;49(5):1601526. doi: 10.1183/13993003.01526-2016. Print 2017 May. PMID 28461290
- [Result] Cottini M, Lombardi C, Passalacqua G, Bagnasco D, Berti A, Comberiati P, Imeri G, Landi M, Heffler E. Small Airways: The "Silent Zone" of 2021 GINA Report? Front Med (Lausanne). 2022 May 23;9:884679. doi: 10.3389/fmed.2022.884679. eCollection 2022. PMID 35677830